CLINICAL TRIAL: NCT06116019
Title: A Prospective Study on Online Adaptive Radiotherapy (ART) Using the ETHOS Linear Accelerator for Various Tumor Entities and the Feasibility of Integrating Multi-Parametric Patient Data Into the Adaptive Workflow
Brief Title: Online Adaptive Radiotherapy Using a Novel Linear Accelerator (ETHOS)
Acronym: ART-02
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Goda Kalinauskaite, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: 3000902
Record Dates: First submitted 2023-09-22; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer; Head and Neck Cancer; NSCLC; SCLC; Esophageal Cancer; Bladder Cancer; Rectum Cancer; Cervix Cancer; Other Carcinoma
Keywords: online adaptive radiation therapy; ART; cone beam CT; ePROMS
MeSH Terms: conditions — Prostatic Neoplasms; Head and Neck Neoplasms; Esophageal Neoplasms; Urinary Bladder Neoplasms; Rectal Neoplasms; Uterine Cervical Neoplasms; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Radiation: Online adaptive radiation therapy — Daily cone-beam CT based online adaptive radiation therapy

SUMMARY:
The study focuses on the scientific and clinical evaluation of online adaptive radiotherapy (ART) using the Varian/SHS ETHOS treatment system. In this study, radiation treatment plans are dynamically adjusted on a daily basis over several weeks of therapy to account for anatomical shifts in either the tumour or adjacent normal tissue - a capability that has been difficult to achieve due to technical limitations. With the ETHOS accelerator, such real-time adjustments can be made based on cone beam computed tomography (CBCT). This is a prospective observational study with the primary objective of investigating the feasibility and acceptability of performing ART with ETHOS for different tumour entities. The study will also evaluate the feasibility of integrating multi-parametric data sets into the ART workflow, such as standardised electronic feedback on treatment toxicity from both patients (ePROMS) and physicians (ePRT).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* All tumor entities with an indication for radiotherapy and/or chemoradiotherapy
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Patients who are not capable of giving consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years, diagnosed with malignancies that have an indication for radiation therapy, with or without concurrent chemotherapy, and who are receiving online adaptive radiation therapy at the Department of Radiation Oncology at Charité.
Sampling Method: Probability Sample
Enrollment: 649 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2026-10-09 (Estimated); Study Completion 2027-10-09 (Estimated)

PRIMARY OUTCOMES:
Number of Successfully Completed Adaptive Radiotherapy Sessions in Patients with Various Tumor Entities | Throughout the treatment period, up to 6 weeks.
  This measure evaluates the success rate of adaptive radiotherapy sessions with ETHOS across different tumor types. It measures the total count of adaptive treatment sessions that were completed without interruption or complication for each patient.

SECONDARY OUTCOMES:
Number of Adaptive Radiotherapy Sessions with Dosimetric Benefits to Target Coverage in Patients with Various Tumor Entities | Throughout the treatment period, up to 6 weeks.
  This measure quantifies the adaptive treatment sessions for which a dosimetric advantage for target coverage is detected in patients undergoing adaptive radiotherapy across different tumor types.
Number of Adaptive Radiotherapy Sessions with Dosimetric Benefits to Organs at Risk in Patients with Various Tumor Entities | Throughout the treatment period, up to 6 weeks.
  This measure quantifies the adaptive treatment sessions for which a dosimetric advantage for organs at risk is detected in patients undergoing adaptive radiotherapy across different tumor types.
Number of Adaptive Radiotherapy Sessions with Dosimetric Benefit to Organs at Risk Following ePROMs and ePRT-based Plan Adjustments in Patients with Various Tumor Entities | Throughout the treatment period, up to 6 weeks.
  This measure quantifies the adaptive treatment sessions for which in silico analysis identifies a potential dosimetric advantage to organs at risk following ePROMs and ePRT-based plan adjustments.
Patient Reported Toxicity | 2 years
  Frequency and severity of treatment-related toxicities in patients as scored using the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (NCI-PRO-CTCAE)
Physician Reproted Toxicity | 2 years
  Frequency and severity of treatment-related toxicities in patients as scored using the the Common Terminology Criteria for Adverse Events (CTCAE)
Impact of Adaptive Radiotherapy on Patient Quality of Life Assessed by EORTC QLQ-C30 | 2 years
  This measure evaluates the quality of life of patients undergoing adaptive radiotherapy using the EORTC QLQ-C30 scale.
Fatigue Levels in Patients Undergoing Adaptive Radiotherapy Assessed by FACIT-F | 2 years
  This measure quantifies the fatigue experienced by patients undergoing adaptive radiotherapy as determined by the FACIT-F scale.
Local Control | 2 years
  Freedom from local progression after adaptive radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin, Berlin, Germany